CLINICAL TRIAL: NCT03021278
Title: Lumbar Tactile Acuity in Experimentally Induced Acute Low Back Pain
Brief Title: Tactile Acuity in Experimentally Induced Acute Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Jerzy Kukuczka Academy of Physical Education in Katowice (Other)
Collaborators: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Wacław Adamczyk, PhD candidate, The Jerzy Kukuczka Academy of Physical Education in Katowice
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 8/2016
Record Dates: First submitted 2017-01-09; First posted 2017-01-13 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Acute Pain; Low Back Pain
Keywords: Tactile acuity; Chronic pain; Two-point discrimination; Point-to-point test; Two-point estimation; Body image
MeSH Terms: conditions — Acute Pain; Low Back Pain; Chronic Pain | interventions — Sodium Chloride; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Saline Injection (Experimental): In the saline injection group, low back pain will be induced via 1.0 ml hypertonic (5% NaCl).
  Interventions: Other: Saline injection
- Sham Injection (Experimental): In the sham injection group, a real needle will be shown to the participants to imitate and produce the anticipation of a pain experience.
  Interventions: Other: Sham injection
- Control Group (No Intervention): The control group will not receive any kind of pain or pinprick sensation.

INTERVENTIONS:
Other: Saline injection — In the saline injection group, low back pain will be induced via 1.0 ml hypertonic (5% NaCl) saline bolus injection which is a commonly used model of acute low back pain. Saline will be injected into the right (or left) lumbar longissimus muscle 50 mm lateral to the spinous process just above (5 mm) previously marked point. Injections will be performed by a physician under ultrasound imaging guidance to ensure that each single injection will be equally placed at a depth of 30 mm. The side for the pain induction will be randomised across subjects. The place of needle insertion and corresponding point on the opposite side of the body will be covered by placing a small piece of adhesive plaster.
  Other Names: Experimental pain
  Arms: Saline Injection
Other: Sham injection — In the sham-injection group (placebo comparator), a real needle will be shown to the participants to imitate and produce the anticipation of a pain experience. A pinprick sensation will be produced by a weighted stimulus applied perpendicularly to the skin just above without piercing the skin. A stimulus of 512 mN will be used to produce a pinprick sensation and activation of cutaneous nociceptors. Adhesive tapes covering stimulation points will also be provided.
  Other Names: Sham pain
  Arms: Sham Injection

SUMMARY:
The purpose of this study is to determine whether experimentally induced acute low back pain might lead to alteration in lumbar tactile acuity measured in region affected by pain compared to pain-free side and pain-free controls.

DETAILED DESCRIPTION:
Healthy male participants will be recruited at the Academy of Physical Education in Katowice. Each participant will be assessed only once. All participants will be asked to provide written informed consent for participation prior to the experimental procedure and will be naïve to the experimental hypothesis. The plan for this research project has been previously approved by the local bioethical committee.

Between-subject (real-injection, sham-injection and control group) and within-subject (assessment 1 versus assessment 2 and 3) design will be used for the purpose of this experiment. After the screening procedure and preparation phase, participants will be randomly assigned to one of three groups: control, saline injection or sham-injection. Groups will differ only in terms of the specific manipulation: the experimental group will receive intra-muscular saline injection, the sham-injection group will be stimulated by pinprick sensation produced by a PinPrick device. No manipulation will take place in the control group allowing to control for the learning effect. In fact, participants will be informed that the study includes only two branches so they can be assigned either to the group with pain evoked as a result of an injection or to the control group without any noxious stimuli. Not revealing the sham-injection condition will allow for comparison between nociceptive (injection) and non-nociceptive (sham-injection) condition.

Because no previous studies have investigated tactile acuity changes in acute low back pain, the sample size calculation was based on the data from our own systematic review and meta-analysis (Adamczyk et al., under review) and previous cross-sectional data among healthy controls (Adamczyk et al., 2016). Based on reported mean difference of 9.49mm between chronic low back pain patients and healthy controls and standard deviation of 9.90mm, a total sample size of 57 participants (19 per group) is required to detect a significant effect. Power calculation was performed for specific planned-comparison tests that were described in detailed under 'statistical analysis' section below. Calculation was performed in G*Power (G*Power 3.1.9.2 statistical software) with the alpha level set at =0.05 and 80% power.

Baseline differences in descriptive statistics will be analysed by one-way analysis of variance (ANOVA) with 'group' as the between-subject factor. Further statistical comparisons will be performed using a repeated-measures ANOVA design, with 'group' (real-injection, sham-injection, and control group) as between-subject factor and repeated measures (assessment 1, 2 and 3) as a within-subject factor. In order to test hypothesis on tactile acuity alteration during pain induction, F-tests will be followed by planned comparisons on data from assessment 1 versus assessment 2 in experimental group. To determine whether the magnitude of tactile acuity alteration has differed between the groups, planned comparisons will be performed on the difference in tactile acuity (assessment 1 vs. assessment 2) between real-injection and sham-injection group and between real-injection and control group. Bonferroni correction will be used for multiple planned comparisons. Forward, stepwise multiple regression will be performed to determine the degree to which tactile acuity change is predicted by either pain intensity or the size of its distribution. All the analyses will be conducted using the STATISTICA data analysis software, version 12 (StatSoft Inc., Tulsa, OK, USA). The level of significance will be set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Only participants with similar mechanical detection threshold (MDT) on both sides of the spine will be included.

Exclusion Criteria:

* sex: female
* age < 18 or > 35 years
* laterality: left-handed
* current pain experience
* episodes of back pain lasting more than 24 hours within the previous one-month period
* history of chronic pain, i.e. pain lasting more than one-month
* comorbidities affecting the nervous system
* cardio-vascular diseases
* psychiatric illnesses
* any disease requiring systematic drug consumption.
* diagnosed hypersensitive reaction to saline solution

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2017-01; Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Lumbar tactile acuity measured by two-point discrimination test (TPD). | Measured an average 3 minutes after manipulation (e.g. saline injection).
  Mechanical callipers will be delicately applied to the pre-marked axis until the very first blanching of the skin. Testing will be commenced with 0 mm between the two calliper's tips, and then the distance between them will be gradually increased until participants will able to verbally report that two points had been touched instead of one. Subsequently, the descending sequence will be applied until the perception of the two points disappeared.

SECONDARY OUTCOMES:
Pain intensity measured behaviourally on a Numerical Rating Scale (NRS). | Pain intensity will be measured just after saline/sham injection and every 30 seconds after this time point up until 12 minutes.
  The scale for pain intensity ratings will range from 0 = "no pain" to 10 = "the worst pain imaginable"
Distribution of pain measured by estimating the diameter of the circle representing area affected by pain. Greater circle (diameter) will refer to the greater distribution of pain (larger body surface affected). | Pain distribution will be measured just after saline/sham injection and every 30 seconds after this time point up until 12 minutes.
  Greater circle (diameter in cm) will refer to the greater distribution of pain (larger body surface affected).
Fear of pain measured on a Numerical Rating Scale (NRS). | Fear of pain measured only at baseline
  Fear of pain will be rated on a scale ranging from 0 = "not at all" to 10 = "very much".
Lumbar tactile acuity measured by point-to-point test (PTP). | PTP measured at baseline (1), an average 3 minutes after manipulation (2) (e.g. saline injection) and 12 minutes after manipulation (3)
  To perform PTP, participants will be asked to maintain a pen perpendicularly to the surface around the sacrum. Then, the examiner will lightly touch one of the pre-marked point at the participants' back. The participants will be instructed to touch the point that was stimulated by assessor. To analyse PTP, the distance between pre-marked point and points indicated by the participants will be measured with callipers.
Lumbar tactile acuity measured by two-point estimation test (TPE) | PTP measured at baseline (1), an average 3 minutes after manipulation (2) (e.g. saline injection) and 12 minutes after manipulation (3)
  For the two-point estimation test, assessor will apply one tactile stimulus until the very first blanching of the skin, with a 120 mm horizontal separation between the callipers' tips. Subsequently to the tactile stimulation, patients will be asked to manually indicate with their callipers the distance they have perceived (TPE score).

OTHER OUTCOMES:
Fear of Pain Questionnaire (FPQ-III). | Measured only at baseline
  FPQ-III consists of three subscales measuring: minor pain, severe pain, and medical pain. Each subscale contains 10 items. The total score has a range 30-150. A higher score indicates greater fear of pain.
Pain Catastrophizing Scale (PCS). | Measured only at baseline
  The PCS scale includes 13 items creating three subscales: magnification, rumination and helplessness. All three scales measure a tendency to exaggerate and misinterpret threatening situations.

CONTACTS AND LOCATIONS:
Overall Officials: Wacław M Adamczyk, Msc, Principal Investigator — The Jerzy Kukuczka Academy of Physical Education
Locations (1):
- The Jerzy Kukuczka Academy of Physical Education, Katowice, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adamczyk W, Slugocka A, Saulicz O, Saulicz E. The point-to-point test: A new diagnostic tool for measuring lumbar tactile acuity? Inter and intra-examiner reliability study of pain-free subjects. Man Ther. 2016 Apr;22:220-6. doi: 10.1016/j.math.2015.12.012. Epub 2016 Jan 2. PMID 26797175
- [Background] Catley MJ, O'Connell NE, Berryman C, Ayhan FF, Moseley GL. Is tactile acuity altered in people with chronic pain? a systematic review and meta-analysis. J Pain. 2014 Oct;15(10):985-1000. doi: 10.1016/j.jpain.2014.06.009. Epub 2014 Jun 28. PMID 24983492
- [Background] Tsao H, Tucker KJ, Coppieters MW, Hodges PW. Experimentally induced low back pain from hypertonic saline injections into lumbar interspinous ligament and erector spinae muscle. Pain. 2010 Jul;150(1):167-172. doi: 10.1016/j.pain.2010.04.023. Epub 2010 May 26. PMID 20510516
- [Background] Wand BM, Di Pietro F, George P, O'Connell NE. Tactile thresholds are preserved yet complex sensory function is impaired over the lumbar spine of chronic non-specific low back pain patients: a preliminary investigation. Physiotherapy. 2010 Dec;96(4):317-23. doi: 10.1016/j.physio.2010.02.005. PMID 21056167
- [Derived] Adamczyk WM, Saulicz O, Saulicz E, Luedtke K. Tactile acuity (dys)function in acute nociceptive low back pain: a double-blind experiment. Pain. 2018 Mar;159(3):427-436. doi: 10.1097/j.pain.0000000000001110. PMID 29140929
- See also: Protocol of the meta-analysis on lumbar tactile acuity in patients with low back pain and healthy controls — https://www.crd.york.ac.uk/prospero/display_record.asp?ID=CRD42016037217